CLINICAL TRIAL: NCT05812729
Title: A Randomized Controlled Study to Evaluate the Feasibility and Efficacy of an Online Resilience Intervention in the General Population ("resiLIR Basic")
Brief Title: "resiLIR Basic": A Psychological Online Intervention to Enhance Resilience in the General Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leibniz-Institut für Resilienzforschung (LIR) gGmbH (Other)
Collaborators: European Regional Development Fund (Other); Ministry of Science and Health of Rhineland-Palatinate, Germany (Unknown); Fraunhofer Institute for Industrial Mathematics ITWM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01_resiLIR_basic
Record Dates: First submitted 2023-02-24; First posted 2023-04-14 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Resilience

STUDY DESIGN:
Intervention Model Description: Waitlist-control design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will receive access to the 6-week online resilience intervention "resiLIR Basic" consisting of 8 modules of about 45-60 minutes addressing evidence-based resilience factors, such as optimism or sense of coherence.
  Interventions: Behavioral: resiLIR Basic
- Waitlist control group (No Intervention): Participants will receive the intervention after the first follow-up assessment (3 months after post-assessment).

INTERVENTIONS:
Behavioral: resiLIR Basic — Each module contains psychoeducational elements as well as practical exercises.
  Week 1: Introduction + "Stress and resilience"
  Week 2: "Optimism"
  Week 3: "Mindfulness"
  Week 4: "Sense of coherence and values"
  Week 5: "Acceptance"
  Week 6: "Self-compassion" + Conclusion
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to examine the developed online resilience intervention "resiLIR Basic" for the general population.

Participants will receive a 6-week online intervention addressing resilience and stress as well as different resilience factors. The main question is whether the intervention is effective in increasing psychological resilience.

DETAILED DESCRIPTION:
Background: Acute and chronic stress in everyday life plays an essential role in the onset and development of several physical and mental health conditions. The ability to maintain or return to mental health during stress exposure is characterized as resilience. Especially the COVID-19 pandemic emphasized the role of resilience for mental health and pointed to the importance of easily accessible and flexible interventions to improve resilience in the general population.

Objectives: The aim of the study therefore is to examine the feasibility and efficacy of a newly developed online intervention to foster resilience in the general population.

Methods: In a waitlist control design, 240 adults will participate in the 6-week resilience intervention "resiLIR Basic". This online intervention consists of 8 modules of about 45-60 minutes length using psycho-educational elements and practical exercises to address evidence-based resilience factors, such as optimism or sense of coherence. Participants will complete online surveys on resilience, mental health, and several resilience factors pre-, during and post-intervention as well as 3, 6 and 12 months after completion as follow-up assessments.

Implications: The study will contribute to an evidence-based and easily accessible supply of resilience interventions supporting health promotion and stress prevention in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Fluent in German language
* Have access to an internet-enabled device with a large screen (tablet / laptop / computer).
* as well as that they can use at least once a week for 45 min to 1.5 hours during the study period

Exclusion Criteria:

* Acute mental health crisis (e.g., suicidality)
* Psychiatric/psychotherapeutic treatment
* Neurodegenerative disease(s)
* Diagnosis of schizophrenia or other psychotic disorders, bipolar disorder, post-traumatic stress disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Change of Resilience measured with stressor reactivity score (Kalisch et al., 2015, 2021) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Stressor reactivity score (Kalisch et al., 2015, 2021): Stressor reactivity can be approximated by relating self-reported mental-health problems to the corresponding stressor exposure within the same timeframe (for scales for mental health problems and stressor exposure, see secondary outcomes). The stressor reactivity (SR) score will be computed as an individual score against normal stressor reactivity (see Kalisch et al., 2021), where normal stressor reactivity is the regression line of average mental health problems against average stressor exposure across all time points in the trial population and one's individual SR score at any time point is the distance to the regression line. The inverse of the SR score is considered an approximative index of outcome-based resilience. Therefore, a lower SR score indicates higher resilience. Change calculated between time points named in time frame, for details, see statistical analysis plan.

SECONDARY OUTCOMES:
Change of Resilience as measured by the Brief Resilience Scale (BRS; Chmitorz et al., 2018) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Brief Resilience Scale (BRS; Chmitorz et al., 2018): Participants rate 6 items on a scale from 1 to 5. Items 2, 4 and 6 are inverted; scale mean is formed. Higher scores indicate higher resilience. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Mental Health measured by the General Health Questionnaire (GHQ-12; Schrnitz et al., 1999) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  General Health Questionnaire (GHQ-12; Schrnitz et al., 1999): Participants rate 12 items on a scale from 0 to 3. Items 14, 15, 10, 16, 18 and 19 are inverted; sum score is formed. Higher scores indicate lower mental health. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Optimism measured with Optimism-Pessimism-Scale (SOP-2; Kemper et al., 2014) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Optimism-Pessimism-Scale (SOP-2; Kemper et al., 2014): Participants rate different items on a scale from 1 to 7. Item 2 is inverted, scale mean is formed. Higher scores indicate higher optimism. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Mindfulness measured with Mindful Attention and Awareness Scale (MAAS-Short; Höfling et al., 2011) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Mindful Attention and Awareness Scale (MAAS-Short; Höfling et al., 2011) Participants rate different items on a scale from 1 to 6. Items 1, 2, 3, 4 and 5 are inverted; scale mean is formed. Higher scores indicate higher mindfulness. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Sense of Coherence measured by Sense of Coherence Scale-29 (SOC-29; Singer et al., 2007) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Sense of Coherence Scale-29 (SOC-29; Singer et al., 2007): Participants rate different items on a scale from 1 to 7. Item 2, 5, 6, 7, 8, 12, 14, 15, 17, 21, 24 and 28 are inverted, scale mean is formed. Higher scores indicate higher sense of coherence. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Meaning and Purpose measured by Subscale of Comprehensive Inventory of Thriving (CIT; Hausler et al., 2017) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Subscale of Comprehensive Inventory of Thriving (CIT; Hausler et al., 2017): Participants rate different items on a scale from 1 to 5. Scale mean is formed. Higher scores indicate higher meaning. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Positive Reappraisal measured with Subscale of Cognitive Emotion Regulation Questionnaire (CERQ; Loch et al., 2011) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Subscale of Cognitive Emotion Regulation Questionnaire (CERQ; Loch et al., 2011): Participants rate different items on a scale from 1 to 6. Scale mean is formed. Higher scores indicate higher positive reappraisal. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Acceptance measured with Subscale of Cognitive Emotion Regulation Questionnaire (CERQ; Loch et al., 2011) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Subscale of Cognitive Emotion Regulation Questionnaire (CERQ; Loch et al., 2011) Participants rate different items on a scale from 1 to 6. Scale mean is formed. Higher scores indicate higher acceptance. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Self Compassion measured with Self-Compassion Scale Deutsch (SCS-D; Hupfeld & Ruffieux, 2011) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Self-Compassion Scale Deutsch (SCS-D; Hupfeld & Ruffieux, 2011): Participants rate different items on a scale from 1 to 5. Items 1, 2, 4, 6, 8, 11, 13, 16, 18, 20, 21, 24 and 25 are inverted; Scale mean is formed. Higher scores indicate higher self compassion. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Perceived Stress measured with Perceived Stress Scale (PSS-2+2; Schäfer et al., in preparation) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Perceived Stress Scale (PSS-2+2; Schäfer et al., in preparation): Participants rate different items on a scale from 1 to 5. Items 1 and 2 are inverted; scale mean is formed. Higher scores indicate higher stress. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Depression measured with Patient Health Questionnaire-9 (PHQ-9; Löwe et al., 2002) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Patient Health Questionnaire-9 (PHQ-9; Löwe et al., 2002): Participants rate 9 items on a scale from 0 to 3. Sum score is formed. Higher scores indicate higher depression. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Anxiety measured with Generalized Anxiety Disorder-7 (GAD-7; Löwe et al., 2002) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Generalized Anxiety Disorder-7 (GAD-7; Löwe et al., 2002): Participants rate 7 items on a scale from 0 to 3. Sum score is formed. Higher scores indicate higher anxiety. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Well-being measured with WHO-5 Well-Being Index (Brähler et al., 2007) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  WHO-5 Well-Being Index (Brähler et al., 2007): Participants rate 5 items on a scale from 1 to 6. Sum score is formed. Higher scores indicate higher well-being. Change calculated between time points named in time frame, for details, see statistical analysis plan.
Change of Self-Efficacy measured with German Version of Self-Efficacy Short Scale (ASKU; Beierlein et al., 2014) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  German Version of Self-Efficacy Short Scale (ASKU; Beierlein et al., 2014): Participants rate different items on a scale from 1 to 5. Scale mean is formed. Higher scores indicate higher self-efficacy. Change calculated between time points named in time frame.
Change of Positive Appraisal Style (procedural aspects) measured with Positive Appraisal Style Content (PASS-process; no publication, pre-version in Petri-Romao et al., 2021) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Positive Appraisal Style Content (PASS-process; no publication, pre-version in Petri-Romao et al., 2021): Participants rate different items on a scale from 1 to 5. Scale mean is formed. Higher scores indicate higher positive appraisal (procedural aspects). Change calculated between time points named in time frame.
Change of Positive Appraisal Style (content aspects) measured with Positive Appraisal Style Content (PASS-content; no publication, pre-version in Petri-Romao et al., 2021) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Positive Appraisal Style Content (PASS-content; no publication, pre-version in Petri-Romao et al., 2021): Participants rate different items on a scale from 1 to 4. Scale mean is formed. Higher scores indicate higher positive appraisal (content aspects). Change calculated between time points named in time frame.
Change of Social Support measured with Oslo Social Support Scale (OSS-3; Kocalevent et al., 2018) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Oslo Social Support Scale (OSS-3; Kocalevent et al., 2018): Participants rate different items on a scale from 1 to 4/ 1 to 5. Sum score is formed. Higher scores indicate higher social support. Change calculated between time points named in time frame.
Change of Internal and External Locus of Control measured with Internal-External Locus of Control Short Scale-4 (IE-4; Kovaleva et al., 2014) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Internal-External Locus of Control Short Scale-4 (IE-4; Kovaleva et al., 2014): Participants rate different items on two subscales from 1 to 5. Scale mean for each subscale is formed. Higher scores on the first subscale indicate higher internal locus of control, higher scores on the second subscale indicate higher external locus of control. Change calculated between time points named in time frame.
Change of Coping measured with Coping Orientation to Problems Experienced Inventory (Brief-COPE; Knoll et al., 2005) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Coping Orientation to Problems Experienced Inventory (Brief-COPE; Knoll et al., 2005): Participants rate different items on two subscales from 1 to 4. Scale mean for each subscale is formed. Higher scores on the first subscale indicate higher adaptive coping, higher scores on the second subscale indicate higher maladaptive coping. Change calculated between time points named in time frame.
Change of Self-Esteem German Single-Item Self-Esteem Scale (G-SISE; Brailovskaia & Margraf, 2020) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  German Single-Item Self-Esteem Scale (G-SISE; Brailovskaia & Margraf, 2020):
  Participants rate one item on a scale from 1 to 5. Higher scores indicate higher self-esteem. Change calculated between time points named in time frame.
Change of Positive Affect measured with Subscale of Positive and Negative Affect Schedule (PANAS; Breyer & Bluemke, 2016) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Subscale of Positive and Negative Affect Schedule (PANAS; Breyer & Bluemke, 2016) Participants rate 10 items on a scale from 1 to 5. Scale mean is formed. Higher scores indicate higher positive affect. Change calculated between time points named in time frame.
Change of Satisfaction with Life measured with Satisfaction with Life Scale (SWLS; Janke & Glöckner-Rist, 2012) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Satisfaction with Life Scale (SWLS; Janke & Glöckner-Rist, 2012):
  Participants rate 5 items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher satisfaction with life. Change calculated between time points named in time frame.
Change of Functioning measured with World Health Organization Disability Assessment Schedule (WHODAS 2.0; Üstün et al., 2010) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  World Health Organization Disability Assessment Schedule (WHODAS 2.0; Üstün et al., 2010):
  Participants rate 12 items on a scale from 1 to 5. Sum score is formed. Higher scores indicate lower functionality. Change calculated between time points named in time frame.
Change of Coping Flexibility measured with Coping Flexibility Questionnaire Revised (CFQ-R; Kato, 2020) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Coping Flexibility Questionnaire Revised (CFQ-R; Kato, 2020):
  Participants rate 12 items on a scale from 1 to 4. There are three sub scales. Scale mean is formed, respectively. Higher scores indicate higher flexibility. Change calculated between time points named in time frame.
Satisfaction with Intervention (only intervention group) measured with Client Satisfaction Questionnaire-Intervention (CSQ-I; Boß et al., 2016) | 6-8 weeks (post)
  Client Satisfaction Questionnaire-Intervention (CSQ-I; Boß et al., 2016):
  Participants rate 8 items on a scale from 1 to 4. Scale mean is formed. Higher scores indicate higher client satisfaction.
Adverse effects (only intervention group) measured with Inventory of Negative Effects of Psychotherapy for Online-Interventions (INEP-ON; Ladwig et al., 2014) | 6-8 weeks (post)
  Inventory of Negative Effects of Psychotherapy for Online-Interventions (INEP-ON; Ladwig et al., 2014): Participants rate in total 23 items. Of these, items 1 to 11 are rated on a 7-point scale ranging from 3 (positive outcome, like "better" or "supportive") to -3 (negative outcome, like "worse" or "disturbing"); items 12 to 21 are rated on a 4-point scale ranging from 0 (fully disagree) to 3 (fully agree) and then rated if a possible change is attributed to the intervention or life circumstances. Items 22 and 23 are also rated on a 4-point scale ranging from 0 (fully disagree) to 3 (fully agree).
  We are not sure whether the questionnaire can be evaluated with a sum score or mean, we have contacted the author about it to receive instructions.
Relationship to Intervention (only intervention group) measured with Mobile Agnew Relationship Measure (mARM; von Wulffen et al., 2022): | 6-8 weeks (post)
  Mobile Agnew Relationship Measure (mARM; von Wulffen et al., 2022): Participants rate 24 items on a scale from 1 to 7. Items 4, 8, 16, and 18 are reverse coded. There are 5 sub scales. Scale mean is formed, respectively. Higher scores indicate higher bond/ confidence/ openness/ relationship/ client initiative.

OTHER OUTCOMES:
Change of Self-care measured with Hamburg Self-Care Survey (Harfst et al., 2009) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Hamburg Self-Care Survey (Harfst et al., 2009): Participants rate 12 items on a scale from 1 to 5. Scale mean is formed. Higher scores indicate higher self-care. Change calculated between time points named in time frame.
Attitudes towards Psychological Online Interventions measured with Attitudes towards Psychological Online Interventions Questionnaire (APOI; Schröder et al., 2015) | baseline (pre)
  Attitudes towards Psychological Online Interventions Questionnaire (APOI; Schröder et al., 2015):
  Participants rate 16 items on a scale from 1 to 7. There are four sub scales (Scepticism and perception of Risks, Confidence in Effectiveness, Technologization Threat, Anonymity Benefits), scale mean is formed, respectively. Higher scores indicate higher Scepticism, etc..
Personality measured with Big Five Inventory-10 (BFI-10; Rammstedt et al., 2017) | baseline (pre)
  Big Five Inventory-10 (BFI-10; Rammstedt et al., 2017):
  Participants rate 10 items on a scale from 1 to 5. There are five sub scales (Extraversion, Openness, Neuroticism, Agreeableness, Conscientiousness). Scale mean is formed, respectively. Higher scores indicate higher Extraversion, etc.
Sociodemographic Variables | baseline (pre)
  Single Items: age, sex, education
Socioeconomic Variables | baseline (pre)
  number of people living in household, household net income, individual net income
Change of Belief Towards Mental Illness measured with Belief Towards Mental Illness Scale (Hirai & Clum, 2018) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Belief Towards Mental Illness Scale (Hirai & Clum, 2018):
  Participants rate 21 items on a scale from 1 to 6. There are three sub scales (Dangerousness, Poor social and interpersonal skills, Incurability). Scale mean is formed, respectively. Higher scores indicate higher Dangerousness, etc.Change calculated between time points named in time frame.
Change of Help-seeking Behavior measured with General Help Seeking Scale (Rickwood et al., 2005) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  General Help Seeking Scale (Rickwood et al., 2005):
  Participants rate 15 items on a scale from 1 to 4. There are three sub scales (level of intention for seeking informal help, level of intention for seeking formal help, level of intention to seek help from no-one). Scale mean is formed, respectively. Higher scores indicate higher level of intention for seeking informal help, etc. Change calculated between time points named in time frame.
Change of Attitudes towards Help-seeking Behavior measured with Attitudes Toward Seeking Professional Psychological Help (Kessler et al., 2015) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Attitudes Toward Seeking Professional Psychological Help (Kessler et al., 2015) Participants rate 24 items on a scale from 1 to 5. Items 1, 3, 4, 6, 7, 9, 11, 12, 14, 16, 17, 18, 20, 21 and 24 are inverted. There are three sub scales (Psychological Openness, Help-Seeking Propensity, Indifference to stigma). Scale mean is formed, respectively. Higher scores indicate higher level of Psychological Openness, etc. Change calculated between time points named in time frame.
Change of Mental Health Literacy measured with Mental Health Literacy Questionnaire (Dias et al., 2018) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Mental Health Literacy Questionnaire (Dias et al., 2018):
  Participants rate 29 items on a scale from 1 to 5. Items 6, 10, 13, 15, 21 and 23 are invertedSum score is formed. Higher scores indicate higher health literacy.Change calculated between time points named in time frame.
Change of Mental Health Literacy measured with Mental Health Literacy Scale (O'Connor & Casey, 2015) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Mental Health Literacy Scale (O'Connor & Casey, 2015):
  Participants rate 35 items on a scale from 1 to 4/5. Items 10, 12, 15, 20, 21, 22, 23, 24, 25, 26, 27, 28 are inverted. Sum score is formed. Higher scores indicate higher health literacy. Change calculated between time points named in time frame.
Change of Mental Health Literacy measured with Mental Health Knowledge Schedule (Evans-Lacko et al., 2010) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Mental Health Knowledge Schedule (Evans-Lacko et al., 2010) Participants rate 6 items on a scale from 1 to 6. Sum score is formed where 6 (don't know) is equalized to a score of 3. Higher scores indicate higher health literacy. Change calculated between time points named in time frame.
Change of Mental Health Literacy measured with Health Literacy Survey EU 16 (Jordan & Hoebel, 2015) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Health Literacy Survey EU 16 (Jordan & Hoebel, 2015) Participants rate 16 items on a scale from 1 to 4. Sum score is formed where 1/2 are summed up to a score of 1 and 3/4 are summed up to a score of 0. Higher scores indicate higher health literacy. Change calculated between time points named in time frame.
Change of eMental Health Literacy measured with eHealth Literacy Scale (Soellner et al., 2014) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  eHealth Literacy Scale (Soellner et al., 2014): Participants rate 8 items on a scale from 1 to 5. There are two subscales (Information seeking/ Information appraisal). Scale mean is formed. Higher scores indicate higher information seeking/ information appraisal. Change calculated between time points named in time frame.
Change of Mental Health Literacy measured with Well-being Literacy Scale (Hou et al., 2021): | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Well-being Literacy Scale (Hou et al., 2021): The scale consists of 6 items. Each item is rated on a 7-point Likert scale, from 1 (Strongly disagree) to 7 (Strongly agree). Scale mean is formed. Higher scores indicate higher mental health literacy. Change calculated between time points named in time frame.
Change of Stress measured with STRESS K-10 (Giesinger et al., 2008) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  STRESS K-10 (Giesinger et al., 2008):
  Participants rate 10 items on a scale from 1 to 5. Sum score is formed. Higher scores indicate higher stress. Change calculated between time points named in time frame.
Change of Knowledge of psychosocial care structures measured with Questionnaire to survey knowledge of psychosocial care structures. (Fritz, 2021, in preparation) | baseline (pre), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Questionnaire to survey knowledge of psychosocial care structures. (Fritz, 2021, in preparation) Participants rate 8 items on a scale from 1 to 3 (yes, no, I don't know). Sum score is formed. Higher scores indicate higher knowledge. Change calculated between time points named in time frame.
Occurrence of Stressors within the last week measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | baseline (pre)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020): Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors.
Occurrence of Stressors within the last week measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | 3-4 weeks (intermediate)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020): Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors.
Occurrence of Stressors within the last week measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | baseline (pre), 3-4 weeks (intermediate), 6-8 weeks (post), 3 months (first follow-up), 6 months (second follow-up), 12 months (third follow-up)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020): Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors.
Occurrence of Stressors within the last week measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | 6-8 weeks (post)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020): Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors.
Occurrence of Stressors within the last week measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | 3 months (first follow-up)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020): Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors.
Occurrence of Stressors within the last week measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | 6 months (second follow-up)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020): Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors.
Occurrence of Stressors within the last week measured with Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020) | 12 months (third follow-up)
  Mainz Inventory for Micro Stressors (MIMIS; Chmitorz et al., 2020): Participants rate different items on a scale from 1 to 7. Sum score is formed. Higher scores indicate higher number of stressors.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | baseline (pre)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017): Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | 3-4 weeks (intermediate)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017): Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | 6-8 weeks (post)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017): Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | 3 months (first follow-up)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017): Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | 6 months (second follow-up)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017): Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.
Occurrence of Life Events measured with Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017) | 12 months (third follow-up)
  Life Events Checklist-5 (LEC-5; Krüger-Gottschalk et al., 2017): Participants rate different items on a scale from 1 to 6. Items experienced directly are weighted by a factor of 3, items witnessed weighted with a factor of 2, items learned about or experienced at work are weighted with a factor of 1. Sum score is formed. Higher scores indicate more events experienced with closer proximity to the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Tüscher, Principal Investigator — Leibniz Institute of Resilience Research
Locations (1):
- Leibniz Institute for Resilience Research gGmbH, Mainz, Rhineland-Palatinate, Germany

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT05812729/SAP_000.pdf